CLINICAL TRIAL: NCT02294851
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of Intravenously Administered BMS-986168 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CN002-001
Record Dates: First submitted 2014-11-12; First posted 2014-11-19 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Tauopathies
MeSH Terms: conditions — Tauopathies | interventions — gosuranemab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Ascending dose cohorts (Experimental): Single ascending dose escalation, safety, tolerability, PK, PD and immunogenicity study of BMS-986168 administered by an intravenous infusion in healthy subjects.
  Interventions: Drug: BMS-986168
- Placebo (Placebo Comparator): BMS-986168 Placebo
  Interventions: Drug: BMS-986168 Placebo

INTERVENTIONS:
Drug: BMS-986168
  Other Names: Other Names: BIIB092
  Arms: Single Ascending dose cohorts
Drug: BMS-986168 Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled, single ascending dose escalation, safety, tolerability, PK, PD and immunogenicity study of BMS-986168 administered by an intravenous infusion in healthy subjects.

DETAILED DESCRIPTION:
This study, previously posted by Bristol-Myers Squibb, has transitioned to Biogen under a licensing agreement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, who have no clinically significant deviation from normal in medical history, physical examination, ECGs and clinical laboratory determinations.
* Body Mass Index (BMI) of 18.5-30 kg/m^2, inclusive. BMI=weight (kg)/[height(m)]^2.
* Males and Females, not of child-bearing potential, ages 21 to 65 years, inclusive. Female subjects must have documented proof that they are not of childbearing potential.
* Male subjects must be willing to use effective birth control and refrain from sperm donation during the entire study and for 200 days after dosing has been completed.

Exclusion Criteria:

* Women who are of childbearing potential or breastfeeding.
* Any significant acute or chronic medical illness.
* Any history of cancer within 5 years of enrollment.
* Any major surgery within 4 weeks of study drug administration.
* Donation of blood or serum > 500 mL to a blood bank or in a clinical study (except screening visit) within 3 months of study drug administration.
* Participation in a clinical study (except a screening visit) within 4 weeks (or 5 half lives, whichever is longer), of study drug administration.
* Inability to be venipunctured and/or tolerate venous access.
* Has smoked or used tobacco products within 6 months prior to study drug administration.
* Recent (within 6 months of study drug administration) drug or alcohol abuse as defined in DSM IV, Diagnostic Criteria for Drug and Alcohol Abuse

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as measured by incidence of AEs, serious AEs, AEs leading to discontinuation, and death as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, and physical and neurological examinations. | 8 months
  To evaluate the safety and tolerability of a single intravenous (IV) infusion of BMS-986168 in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - WCCT Global, LLC, Cypress, California
  - Covance Clinical Research Unit Inc., Dallas, Texas